CLINICAL TRIAL: NCT01017315
Title: Efficacy of Baby Talcum in Prevention of Pruritus Assosiated With Cast; a Randomized Controlled Trial
Brief Title: Efficacy of Baby Talcum in Prevention of Pruritus Assosiated With Cast
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Boonsin Tangtrakulwanich, Department of Orthopaedic surgery, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 52-197-11-4-2
Record Dates: First submitted 2009-11-17; First posted 2009-11-20 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Fracture Distal Radius
Keywords: baby talcum; pruritus; cast
MeSH Terms: conditions — Wrist Fractures; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No application of baby talcum (Experimental): control
  Interventions: Drug: Baby talcum

INTERVENTIONS:
Drug: Baby talcum — 50 grams apply locally prior cast application
  Other Names: "Care" brand of baby talcum

SUMMARY:
This study aims to evaluate the efficacy of baby talcum in prevent pruritus after cast application in orthopaedic patients.

The investigators will do a randomized controlled trial in patient with fracture distal end of radius treated conservatively.

Pruritus score and satisfaction will be monitor along the entire course of cast retention.

ELIGIBILITY:
Inclusion Criteria:

* Fracture distal end radius treated conservatively

Exclusion Criteria:

* open fracture
* skin disease and wound under cast area
* Fracture distal end radius needed surgical management
* Allergy to baby talcum

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Pruritus score | 2 years

SECONDARY OUTCOMES:
Satisfaction score | 2 years
Complication rate | 2 years
Number of antihistamine drugs used | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanich, MD.,Ph.D, Principal Investigator — Prince of Songkla University
Locations (1):
- Prince of Songkla university, Hat Yai, Changwat Songkhla, Thailand